CLINICAL TRIAL: NCT07396766
Title: Dissemination of a Breast Reconstruction Decision Tool Through Social Media and Online Communities- AIM1-B
Brief Title: Dissemination of BREASTChoice AIM1-B
Acronym: BREASTChoice
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 24-1553 AIM1-B; R01CA276408 (NIH)
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Breast Neoplasms
Keywords: web-based patient decision aid; BREASTChoice
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breast cancer survivors (Experimental): Breast cancer survivors.
  Interventions: Behavioral: Baseline Questionnaire; Behavioral: Semi structured Interview; Behavioral: Post Survey

INTERVENTIONS:
Behavioral: Baseline Questionnaire — Participants will be screened and share demographic information during screening. If eligible and screened in, the interviewer will send the self-administered pre-survey Decision Quality Index (DQI).
Behavioral: Semi structured Interview — Participants will participate in a semi-structured interview and review of the adapted BREASTChoice tool.
Behavioral: Post Survey — Participants will take the post-survey to assess breast reconstruction decision quality.

SUMMARY:
This registration covers only Aim 1b, which focuses on testing usability. The study will include 20 participants who are breast cancer patients. Participants will be observed using the tool on their mobile devices, and their experience will be evaluated using a "think-aloud" method to capture their thoughts and reactions. Interviews will include open-ended questions about the content and format of the decision aid, with follow-up prompts to gather feedback on design elements (length, order, graphics), comprehension, ease of use, acceptance, and engagement with the tool. Knowledge will be measured using the Decision Quality Instrument before and after using the tool. Results will be analyzed to develop recommendations for the final version of the tool.

DETAILED DESCRIPTION:
This study is part of a larger project that will update and adapt an existing online decision tool called BREASTChoice. The project includes interviews and user testing with breast cancer survivors, interviews with medical experts, and updates to the website design.

Breast reconstruction after a mastectomy is an important part of breast cancer treatment. It can help restore quality of life and body image, which are often affected after surgery. However, many patients, especially those who identify as Black or Hispanic/Latina are not always offered reconstruction. Some patients also lack information about the risks and benefits, leading to choices that may not match their personal preferences.

The BREASTChoice decision aid was created to help patients make informed choices about breast reconstruction. It has been tested in two clinical studies and shown to improve decision quality. Patients and doctors found it helpful and easy to use, but many asked for a version that works better on mobile devices and can be shared with family and friends.

So far, BREASTChoice has mostly been used in clinics and has not reached many people outside of them. To reach more patients, the tool will be adapted for use on social media and online communities, places where many people already go for health information and support.

In the U.S., most adults use social media (about 81%) and search the internet for health information (about 72%). Even most older adults (60%) go online. Breast cancer survivors are especially active in online groups. Early findings show that survivors would use BREASTChoice if it were available through social media.

Following the Designing for Dissemination approach, and in partnership with three cancer survivor organizations and two clinician groups, this project will adapt BREASTChoice and share it through social media and online communities.

ELIGIBILITY:
Inclusions Criteria To participate in this study, a subject must meet all the eligibility criteria outlined below.

* Age ≥ 18 years at the time of consent
* Able to read and speak English.
* Have had surgery, such as a mastectomy or lumpectomy, to remove some or all of their breast or breasts.
* Breast surgery occurred within the past 8 years.
* Breast surgery was due to a diagnosis of breast cancer, ductal carcinoma in situ, or risk of future breast cancer, by participant report.
* Sex was assigned "Female" at birth

Exclusion Criteria

• Individuals with self-reported or observed unstable medical or psychiatric conditions precluding informed consent or participation in the study will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2029-01-20 (Estimated); Study Completion 2029-01-20 (Estimated)

PRIMARY OUTCOMES:
Change in breast reconstruction knowledge | Up to1 week
  This is knowledge based patient-reported outcome measure uses the Breast Cancer Reconstruction Decision Quality Instrument (DQI). DQ is a 9-item patient-reported measure designed to assess how well patients are informed about breast reconstruction options following breast cancer treatment. The instrument consists of multiple-choice questions with factual, correct answers related to breast reconstruction. Decision quality is quantified as a knowledge score, reflecting the extent to which patients understand key information necessary to make informed reconstruction decisions.
  Scores range from 0% to 100%. The total score is calculated by summing the number of correctly answered items and dividing by the total number of questions (9), with higher scores indicating greater knowledge and higher decision quality.

CONTACTS AND LOCATIONS:
Overall Officials: Clara Lee, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- The University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: UNC Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials